CLINICAL TRIAL: NCT03044951
Title: Cryoballoon Versus Irrigated Radiofrequency Ablation in Patients With Paroxysmal Atrial Fibrillation: A Multi-center, Prospective, Randomized, Controlled Study
Brief Title: Comparison of RF and crYoballoon ablatiOn Therapy of AF（CRYO-AF）
Acronym: CRYO-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qi Jin, Clinical Professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DLY201604
Record Dates: First submitted 2017-01-30; First posted 2017-02-07 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cryoablation; irrigated radiofrequency ablation; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cryoballoon ablation (Experimental): patients who accept cryoballoon ablation
  Interventions: Procedure: cryoballoon ablation
- radiofrequency ablation (Active Comparator): patients who accept radiofrequency ablation
  Interventions: Procedure: radiofrequency ablation

INTERVENTIONS:
Procedure: cryoballoon ablation — cryoballoon ablation：pulmonary vein isolation by cryoballoon
  Arms: cryoballoon ablation
Procedure: radiofrequency ablation — radiofrequency ablation: pulmonary vein isolation by radiofrequency energy
  Arms: radiofrequency ablation

SUMMARY:
It's a multi-center, prospective, randomized, controlled clinical trial of cryoballoon versus radiofrequency ablation for paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The hypothesis of this study is that pulmonary vein isolation with cryoballoon ablation is not inferior to radiofrequency ablation with 3D mapping with respect to clinical safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* ECG recording of atrial fibrillation
* first time of ablation
* refractory to at least one anti-arrhythmia drug
* sign informed consent for participation in the study

Exclusion Criteria:

* had ablation before
* serious heart failure
* left atrial diameter>55mm
* Myocardial infarction, heart surgery or coronary intervention in 3 months before the ablation
* Stroke in 6 months before the ablation
* Endocardial thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-11; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy endpoint (time to first documented clinical recurrence after blanking period) | one year
  the time to first documented clinical recurrence after blanking period (month)
Safety endpoint (Any procedure-related complications) | one year
  Any procedure-related complications

SECONDARY OUTCOMES:
Procedure time (min) | one year
  skin to skin
Left atrial time (min) | one year
X-ray time (min) | one year
time to first time cardiovascular hospitalization (month) | one year
QoL changes at 12 months (Units on a Scale) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Wu, Principal Investigator — Ruijin Hospital
Locations (1):
- Shanghai Rui-Jin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Result] Andrade JG, Khairy P, Macle L, Packer DL, Lehmann JW, Holcomb RG, Ruskin JN, Dubuc M. Incidence and significance of early recurrences of atrial fibrillation after cryoballoon ablation: insights from the multicenter Sustained Treatment of Paroxysmal Atrial Fibrillation (STOP AF) Trial. Circ Arrhythm Electrophysiol. 2014 Feb;7(1):69-75. doi: 10.1161/CIRCEP.113.000586. Epub 2014 Jan 19. PMID 24446022